CLINICAL TRIAL: NCT04404803
Title: Motivations and Barriers to Participating in Ophthalmology Research Projects
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: B00366
Record Dates: First submitted 2018-11-22; First posted 2020-05-28 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Eye Diseases
MeSH Terms: conditions — Eye Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — Patients will be asked to complete a questionnaire about the reasons why they agree / decline to take part in research.

SUMMARY:
The primary objective of this project is to understand the reasons why patients agree / disagree to take part in ophthalmology research. This will be done by asking participants to complete a Research Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Over 16 years old
* Willing to participate by completing the questionnaire
* Must be able to speak and read English

Exclusion Criteria:

* Under 16 years of age
* Not willing to complete the questionnaire

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All individuals will be considered for inclusion in this study regardless of age, disability, gender reassignment, marriage and civil partnership, pregnancy and maternity, race, religion and belief, sex, and sexual orientation except where the study inclusion and exclusion criteria explicitly state otherwise.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2019-01-21 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of motivations to participating in ophthalmology research. | 5 years
  Questionnaire
Assessment of barriers in participating in ophthalmology research | 5 years
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Monika Cien, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No